CLINICAL TRIAL: NCT00561808
Title: In-Vitro Maturation of Oocytes From Polycystic Ovarian Patients Undergoing IVF
Acronym: IVM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30/2007
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: PCO/PCOD; IVM; Immature Oocytes
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — In Vitro Oocyte Maturation Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Observational (Experimental)
  Interventions: Other: In-vitro maturation oocytes

INTERVENTIONS:
Other: In-vitro maturation oocytes — Immature oocytes (development stage GV or M1) will be matured in-vitro in IVM culture medium for approximately 28-32 hours. The oocytes will be routinely observed and when they reach maturation (M2) they will be fertilized. The developed embryo will be transferred to the patient 24 hours post-fertilization.

SUMMARY:
Retrieval of immature oocytes from women with polycystic ovaries, their in-vitro maturation, fertilization and embryo transfer can prevent hormonal treatment that can lead to ovarian hyperstimulation. In addition, it can decrease discomfort and side-effects of routine daily administration of hormones and it can be cost-effective. Thirty healthy women with Polycystic Ovarian Syndrome aged 20-35, with BMI 18-30 kg/msq will be included in the study. Their immature oocytes will be retrieved from small follicles without any hormonal treatment. The oocytes will be fertilized post in-vitro maturation. The developed embryros will be transferred to the patients as in a routine IVF cycle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women diagnosed with Polycystic Ovarian Syndrome with BMI 18-30 kg/sqm, aged 20-35

Exclusion Criteria:

* Every one else

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Maturation rate of oocytes, their fertilization rate, cleavage rate and embryo quality. | one year

SECONDARY OUTCOMES:
Implantation rate and successful delivery. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ellenbogen, MD, Study Director — IVF Unit, Hillel Yaffe Medical Center
Locations (1):
- IVF Unit, Hillel Yaffe Medical Center, Hadera, Israel